CLINICAL TRIAL: NCT02037256
Title: A Pilot Study of Peripheral Blood Hematopoietic Stem Cell Mobilization With the Combination of Bortezomib and G-CSF in Multiple Myeloma and Non-Hodgkin's Lymphoma Patients
Brief Title: Bortezomib and Filgrastim to Promote Stem Cell Mobilization in Patients With Non-Hodgkin Lymphoma or Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Divaya Bhutani, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-134; NCI-2012-01173 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-134 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; B-cell Chronic Lymphocytic Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Progressive Hairy Cell Leukemia, Initial Treatment; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage I Small Lymphocytic Lymphoma; Stage II Multiple Myeloma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Untreated Hairy Cell Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Bortezomib; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Treatment (bortezomib and filgrastim) (Experimental): GROUP A: Bortezomib administered in the evening after comploetion of G-CSF collection or on day 6 of mobilization with G-CSF.
  Interventions: Drug: bortezomib; Biological: filgrastim; Procedure: autologous hematopoietic stem cell transplantation
- B Treatment (bortezomib and filgrastim) (Experimental): GROUP B: Bortexomib administered on days 4 & day 7, before administration of filgrastim.
  Interventions: Drug: bortezomib; Biological: filgrastim; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous hematopoietic stem cell transplantation

SUMMARY:
This clinical trial studies peripheral blood hemapoietic stem cell mobilization with the combination of bortezomib and G-CSF (filgrastim) in multiple myeloma and non-Hodgkin lymphoma patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate if addition of Bortezomib to the mobilization protocol will result with an increase in the levels of circulating peripheral blood stem cells (PBSCs) by at least 2-fold in blood and in the apheresis collections in up to 4-days collection protocol.

II. To assess whether time to neutrophil engraftment is 12 days or less, the historical value.

SECONDARY OBJECTIVES:

I. To test for co-mobilization of lymphoma or myeloma cells by bortezomib and G-CSF using real time polymerase chain reaction (PCR) for non-Hodgkin lymphoma (NHL) patients and by flow cytometry (cluster of differentiation [CD]38+/CD138+ cell) for multiple myeloma (MM) patients.

II. To determine the effect of Bortezomib on the extent of mobilization of dendritic cells subsets, plasmacytoid dendritic cell (pDC)1 and pDC2 and DC1/DC2 ratio by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent form before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Diagnosis of B-type NHL or with multiple myeloma and eligible for autologous transplantation
* No more than 3 prior regimens of chemotherapy (Rituximab is not considered chemotherapy) and 4 weeks out of Bortezomib treatment for MM
* Karnofsky performance status of > 50%
* The patient has recovered from all acute toxic effects of prior chemotherapy
* White blood cell (WBC) > 3.0 x 10^9/L
* Absolute neutrophil count > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L
* Serum creatinine =< 2.2
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) less than two times the upper limit of normal (ULN)
* Total bilirubin less than two times the ULN
* Left ventricle ejection fraction > 50% (by normal echocardiogram [ECHO] or multi gated acquisition scan [MUGA] scan)
* Diffusing capacity of the lung for carbon monoxide (DLCO) > 50%
* Forced vital capacity > 50% of predicted
* Negative for human immunodeficiency virus (HIV)
* Female subject is either post-menopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential , agree to use 2 effective methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) from the time of signing the informed consent form through 30 days after the last dose of Bortezomib, or agree to completely abstain from heterosexual intercourse; women of child bearing potential agree to use an approved form of contraception; male subject, even if surgically sterilized (i.e., status post-vasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse for the duration of the study

Exclusion Criteria:

* Patient has a platelet count of < 100x 10^9/L within 14 days before enrollment
* Patient has an absolute neutrophil count of ANC <1.5 x 10^9/L within 14 days before enrollment
* Patient has creatinine of > 2.2 MG/DL within 14 days before enrollment
* Patient has > 1.5 x ULN total bilirubin
* Patient has >= grade 2 peripheral neuropathy within 14 days before enrollment
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Patient has hypersensitivity to Bortezomib, boron or mannitol
* Female subject is pregnant or breast-feeding; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (b-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Participation in clinical trials with other investigational drugs not included in this trial, within 14 days before enrollment and throughout the duration of this trial
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* A co-morbid condition which, in the view of the investigators, renders the patient at high risk for this study
* An acute medical condition resulting from prior chemotherapy
* Brain metastases or carcinomatous meningitis
* Acute infection
* Fever (temp > 38 degrees Celsius [C]/100.4 degrees Fahrenheit [F])
* Patients of child-bearing potential unwilling to implement adequate birth control
* Patients who have deterioration of their clinical status or laboratory parameters between the time of enrollment and transplant (such that they no longer meet entry criteria) may be removed from study at the discretion of the treating physician or principal investigator
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Radiation therapy within 3 weeks before randomization; enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01-21 (Actual); Study Completion 2015-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Divaya Bhutani, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- A. Standard of Care Mobilization: GROUP A: Standard of care mobiliation: Bortezomib (1.3 mg/m2) in the evening after completion of mobilization with G-CSF
- GROUP B: Alternative Mobilization: GROUP B: Bortezomib (1.3 mg/m2) IV on days 4 and 7 (if needed)
Period: Overall Study
Arm/Group | A. Standard of Care Mobilization | GROUP B: Alternative Mobilization
Started | 3 | 20
Completed (1 withdrew consent prior to Velcade infusion 1 removed from protocol prior to Velcade infusioin 1 failed to comply with protocol requirement to come to transplant in 2 months) | 3 | 17
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawn prior to Velcade | 0 | 2

BASELINE CHARACTERISTICS:
Population: Evaluable participants
Groups:
- Arm A: Pts. receive filgrastim SC on days 1-9 & begin apheresis on day 5. Pts. undergo apheresis for up to 2 days, & receive bortezomib intravenously (IV) over 3-5 seconds after target collection is obtained with filgrastim alone or on the 1st day of collection with the Bortezomib plus filgrastim mobilization, prior to receiving the administration of filgrastim. 2nd apheresis will continue until target stem cell dose is reached or for maximum 4 days. Pts. undergo autologous hematopoietic stem cell transplantation after receiving high dose chemotherapy & peripheral blood stem cell (PBSC) infusion following standard of care procedures.
  bortezomib: Given IV
  filgrastim: Given SC
  autologous hematopoietic stem cell transplantation: Under
- Arm B: Pts. receive filgrastim SC on days 1-8 & receive bortezomib IV over 3-5 seconds on days 4 & day 7, before administration of filgrastim. Pts. undergo apheresis on days 5-8
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 3 | 17 | 20
Age, Categorical [Count of Participants; unit: Participants]
  g: <=18 years | 0 | 0 | 0
  g: Between 18 and 65 years | 2 | 13 | 15
  g: >=65 years | 1 | 4 | 5
Age, Continuous [Median (Full Range); unit: years] | 62 [52 to 67] | 56 [40 to 68] | 58 [40 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 1 | 8 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 2 | 14 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 17 | 20

OUTCOME MEASURES:

1. Primary Outcome: >= 2 Fold Increase in Circulating PBSC's
Description: Participants with >= 2 fold increase in circulating PBSC's in blood and in apheresis collections in up to 4-days collection
Time Frame: Up to 6 months
Population: Evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Bortezomib 1.3 mg/m2: Group A: Bortezomib 1.3 mg/m2 in the evening after completion of 5 day mobilization with G-CSF
- Group B Bortezomib 1/3 mg/m2: Group B Bortezomib 1/3 mg/m2 on day 4 of 5 day GCSF mobilizati
Arm/Group | Group A: Bortezomib 1.3 mg/m2 | Group B Bortezomib 1/3 mg/m2
Number analyzed (Participants) | 3 | 17
Participants
  Doubling | 0 | 4
  Less than doubling | 3 | 13

2. Secondary Outcome: Time to Neutrophil Engraftment
Description: Estimated Median Time to Neutrophil Engraftment, ANC 500
Time Frame: Up to 6 months
Population: Evaluable patients
Measure: Median (95% Confidence Interval); unit: days to ANC 500
Groups:
- Arm A Standard of Care Mobilization: G-CSF 16 mcg/kg/day for 9 days; Bortezomib 1.3 mg/m2 IV on day 6. Blood draws and apheresis on days 5-9.
- Arm B Alternative Mobilization: G-CSF16 mcg/kg/day for 8 days; Bortezomib on days 4 and 7. Blood collection on days 4 & 8, apheresis on days 5-8.
Arm/Group | Arm A Standard of Care Mobilization | Arm B Alternative Mobilization
Number analyzed (Participants) | 3 | 17
days to ANC 500 | 12 [12 to NA] — Two few observations to calculate upper limit | 13 [12 to 14]
Statistical Analysis 1: Comparison: Arm B Alternative Mobilization; Median time to engraftment; Test type: Other; percentage = 0.24, 95% CI 2-sided [0.07 to 0.50]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- A Treatment (Bortezomib and Filgrastim): GROUP A Pts. receive filgrastim SC on days 1-8 & receive bortezomib IV over 3-5 seconds on days 4 & day 7, before administration of filgrastim. Pts. undergo apheresis on days 5-8
  bortezomib: Given IV
  filgrastim: Given SC
  autologous hematopoietic stem cell transplantation: Under
- B Treatment (Bortezomib and Filgrastim): Group B Pts receive filgrastim SC on days 1-8 and receive bortezomib IV over 3-5 seconds on days 4 and day 7 before administraioin of filgrastim. Pts undergo apheresis on days 5-8.
Arm/Group | A Treatment (Bortezomib and Filgrastim) | B Treatment (Bortezomib and Filgrastim)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/17
Other Adverse Events (participants affected / at risk) | 6/6 | 17/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Treatment (Bortezomib and Filgrastim) (N=6) | B Treatment (Bortezomib and Filgrastim) (N=17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypertensive crisis (Cardiac disorders) | 0 (0) | 1 (1)
Mucositis (Immune system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypocalcemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Hyperuricemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Low ionized calcioum (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Infection 1 (Infections and infestations) | 1 (1) | 4 (4)
Infection 2 (Infections and infestations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes